CLINICAL TRIAL: NCT07376278
Title: A Prospective Observational Study for the Predictors of Clinical Outcomes of Deep Brain Stimulation in Parkinson's Disease
Brief Title: Predictors of Clinical Outcomes of Deep Brain Stimulation in Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong University of Science and Technology (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other); Hong Kong Center for Neurodegenerative Diseases (Other)
Responsible Party: Principal Investigator, Danise Au, Assistant scientific officer, Hong Kong University of Science and Technology
Other Study IDs: HREP-2024-0289
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Deep Brain Stimulation; PARKINSON DISEASE (Disorder)
Keywords: deep brain stimulation; DBS; Parkinson's disease; multiomic; transcriptomic; proteomic
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, brain tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment: Parkinson's disease patients who have received deep brain stimulation
  Interventions: Procedure: DBS

INTERVENTIONS:
Procedure: DBS — Deep brain stimulation surgery

SUMMARY:
The goal of this observational study is to identify factors in blood that are associated with response to deep brain stimulation (DBS) surgery in patients with Parkinson's disease. The main questions it aims to answer are:

1. What factors in blood (proteins and RNA) are associated with good vs poor response to DBS?
2. Are these factors able to predict response to DBS?
3. How do these factors change before and after DBS?

Blood and leftover brain tissue (which spontaneously adhere to the surgical instruments) will be taken and routine clinical data (including scores from routine assessments) will be collected from consenting participants who undergo DBS.

DETAILED DESCRIPTION:
This is a prospective observational study that investigates the clinical, proteomic, transcriptomic, and genomic profiles that are associated with DBS response with regards to motor symptoms, axial symptoms, non-motor symptoms, change in medications, activities of daily living (ADLs), and quality of life (QOL). The investigators will take blood samples from participants but will not take extra brain tissue; only leftover brain tissue (which is routinely discarded) that spontaneously adheres to surgical instruments will be collected. Study participation will not change the surgical procedure in any way. The investigators also aim to characterize the change in these multiomic profiles before versus after DBS treatment, to evaluate the ability of these multiomic profiles to predict and stratify response to DBS, and to identify modifiable factors to improve response to DBS. Additionally, the investigators will use these multiomic profiles, patient demographics, and clinical presentation to develop a DBS prediction model with advanced explainable AI (XAI) techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of "Clinically Established PD" as defined by the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease (MDS-PD criteria)
2. Referred for DBS according to standard local clinical guidelines 2a. Significant motor complications despite optimized pharmacological treatment 2ai. UPDRS motor score >30/108 in the off-medication state 2aii. Hoehn and Yahr staging >2.5/5 in the off-medication state 2b. Dopamine responsive 2bi. >33% improvement in UPDRS motor score after levodopa administration 2c. Age ≤75 years 2d. No contraindication to surgery or other significant comorbidity with limited life expectancy 2e. No significant psychiatric problems or cognitive impairment 2f. No structural lesions or features suggestive of atypical parkinsonism or other mimickers of idiopathic PD on neuroimaging

Exclusion Criteria:

1. Unwilling to undergo blood sampling for study purposes
2. Evidence of Parkinsonism due to heavy metal exposure
3. History of neurodevelopmental disorder, neurodegenerative disease other than PD, CNS infection, neuroinflammatory disease (e.g. multiple sclerosis, CNS lupus), malignancy within the last 10 years, cerebrovascular accident, HIV infection, systemic autoimmune disease, alcohol dependence or other substance use
4. Unable to pass DBS pre-operative assessment or unwilling to undergo DBS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients of the movement disorder clinic at Queen Elizabeth Hospital Hong Kong
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2036-02-01 (Estimated); Study Completion 2038-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood proteomic profile | From pre-operative to 5 years post-operative
  Plasma proteins measured using high-throughput ultra-sensitive proteomics platform
Blood transcriptomic profile | From pre-operative to 5 years post-operative
  Bulk RNA-sequencing of blood cells
Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | From pre-operative to 5 years post-operative
  Rating scale that measures non-motor experiences of daily living (part I), motor experiences of daily living (part II), motor function via physical examination (part III), and motor complications (part IV)
  Higher scores indicate a worse outcome
  Range:
  Part I: 0-52 Part II: 0-52 Part III: 0-132 Part IV: 0-24
Hoehn and Yahr (H&Y) stage | From pre-operative to 5 years post-operative
  Staging of overall functional disability in Parkinson's disease
  Higher score indicates a worse outcome
  Range: 0-5 Stage 0: No signs of disease Stage 1: Unilateral disease Stage 1.5: Unilateral plus axial involvement Stage 2: Bilateral disease without impairment of balance Stage 2.5: Mild bilateral disease with recovery on pull test Stage 3: Mild to moderate bilateral disease; some postural instability; physically independent Stage 4: Severe disability; still able to walk / stand unassisted Stage 5: Wheelchair bound or bedridden unless aided

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | From pre-operative to 5 years post-operative
  Assessment of cognitive function in 8 domains: attention and concentration, executive functions, memory, language, visuospatial skills, abstraction, calculations, and orientation
  Higher score indicates a better outcome
  Range: 0-30
Non-Motor Symptoms Scale (NMSS) | From pre-operative to 5 years post-operative
  Assessment of symptomatic burden of non-motor symptoms
  Higher score indicates a worse outcome
  Range: 0-360
Parkinson's Disease Sleep Scale - 2 (PDSS-2) | From pre-operative to 5 years post-operative
  Rating scale assessing sleep disorders in PD
  Higher score indicates a worse outcome
  Range: 0-60
Parkinson's Disease Questionnaire - 39 (PDQ-39) | From pre-operative to 5 years post-operative
  39-item self-report questionnaire assessing health-related quality of life in 8 domains: mobility, activities of daily living, emotional wellbeing, stigma, social support, cognition, communication, and bodily discomfort
  Higher score indicates a worse outcome
  Range: 0-100
Depression, Anxiety, and Stress Scale - 21 (DASS-21) | From pre-operative to 5 years post-operative
  Self-report scale measuring depression, anxiety, and stress
  Higher scores indicate a worse outcome
  Range:
  Depression: 0-42 Anxiety: 0-42 Stress: 0-42
Schwab and England Activities of Daily Living Scale (S&E ADL scale) | From pre-operative to 5 years post-operative
  Assessment of ability to accomplish essential activities of daily living
  Higher score indicates a better outcome
  Range: 0-100%

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ip, Principal Investigator — The Hong Kong University of Science and Technology
Locations (1):
- The Hong Kong University of Science and Technology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No